CLINICAL TRIAL: NCT02870647
Title: Sleep Apnea, Arrhythmias and Cardiac Reverse Remodeling in Heart Failure Patients
Acronym: SYNCHRO
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Strategy changes.
Sponsor: LivaNova (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ICSY03
Record Dates: First submitted 2016-07-15; First posted 2016-08-17 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Sleep Breathing Disorders in the Responders to Cardiac Resynchronisation Therapy (CRT)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm study (Other): only 1 arm - no comparison nor randomization in this study
  Interventions: Other: Echocardiographic, polygraphy, electrocardiography measurements and sleep questionnaire

INTERVENTIONS:
Other: Echocardiographic, polygraphy, electrocardiography measurements and sleep questionnaire — each patient is asked to undergo an echocardiographic, polygraphy, electrocardiography measurements, and respond to 2 sleep questionnaires, both at inclusion and after 6 months

SUMMARY:
Prospective, international, non-randomized, multicentre, clinical investigation (phase IV). The aim of the study is to investigate the correlation between HF, severe SBD, and AF in CRT-P patients at 6 months.

DETAILED DESCRIPTION:
The primary objective is to estimate the change in severity of Sleep Breathing Disorders (SBD) in patients with or without reverse remodeling, in de-novo or upgrade implants, after 6 month follow-up.

The main secondary objective is to assess the prevalence, type and evolution of the SBD, co-morbidities and major adverse cardiac events in each subgroup of HF patients (based on the etiology), up to 12 months follow-up period.

Predictors of the clinical outcomes will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patient successfully* implanted (de-novo implant, upgrade or replacement) with a LivaNova CRT-P device, according to the latest applicable CRT guidelines and IFU
* Signed and dated informed consent
* The subject will be available for postoperative follow-up beyond one year

Exclusion Criteria:

* Chronic hypercapnic respiratory failure (under oxygen therapy - that could confound the results of this study)
* Already included in another clinical study that could confound the results of this study
* Not available to attend routine follow-up visits
* Not able to understand the aim of the study and its procedures
* Minor age (according to local regulation)
* Drug / alcohol addiction or abuse
* Known pregnancy
* Under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2019-06 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
The change in severity of SBD (by means of AHI as determined by PG), in the responders to CRT (reverse remodeling, delta LVESV=>15%) compared to the non-responders, at 6-month follow-up after implant (de-novo or upgrade). | 6 months

SECONDARY OUTCOMES:
The main secondary objective is to assess the type of the SBD in each subgroup of HF patients (based on the etiology), up to 12 months follow-up period. | 12 months

CONTACTS AND LOCATIONS:
Locations (3):
- Ospedale Niguarda Ca Granda, Milan, Italy
- Spain (2):
  - Hospital Clinic de Barcelona, Barcelona
  - CHU de Vigo, Vigo